CLINICAL TRIAL: NCT05352724
Title: Randomized, Double Blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy of a Sports Drink on Hydration, Recovery and Glucemia Control After High-intensity Aerobic Exercise
Brief Title: Clinical Trial to Evaluate the Efficacy of a Sport Drink After High-intensity Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioithas SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Elit. Recov
Record Dates: First submitted 2022-04-06; First posted 2022-04-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-04

CONDITIONS: Hydration; Blood Glucose; Sport Recovery; Microbiota

STUDY DESIGN:
Intervention Model Description: The clinical study has a randomized, double-blind, placebo-controlled design. The patients on the list will be randomized to each of the two intervention groups in a 1:1:1 ratio (33% probability for intervention group 1, 33% for intervention group 2 and 33% for the placebo group)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither the patients themselves nor the researchers involved in the study will know the assigned treatment, since these will be coded. The bottles will be labeled with these numbers and will not show distinctive signs of the treatment group. These lists will be kept by the head of the randomization center, and will be hidden from the study staff and participants. For each new inclusion, the researcher will have to contact the randomization center, which will obtain the assigned treatment code.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydration drink A (Experimental): Water with electrolytes and glucose 625 ml 3 times a week for 4 weeks, during exercise
  Interventions: Dietary Supplement: Hydration drink
- Hydration drink B (Active Comparator): Water with electrolytes and calorie-free sweetener 625 ml 3 times a week for 4 weeks, during exercise
  Interventions: Dietary Supplement: Hydration drink
- Hydration drink C (Placebo Comparator): Water with flavoring and coloring 625 ml 3 times a week for 4 weeks, during exercise
  Interventions: Dietary Supplement: Hydration drink

INTERVENTIONS:
Dietary Supplement: Hydration drink — Intake of the different hydrating drinks for 4 weeks 3 times a week during sports practice

SUMMARY:
Although the general effectiveness of carbohydrate/electrolyte-based functional sports drinks on rehydration, recovery and sports performance has been widely demonstrated, there is controversy about the amounts, proportions and components that ensure the effectiveness of these products.

The present study intends to analyze the specific effects of the beverages to be studied on these parameters, taking into account their particular formulation.

Advances in research have allowed us to understand the importance of the intestinal microbiota on health, recovery and performance in sports. The consumption of functional drinks based on carbohydrates and electrolytes as supplementation is a constant in sports environments, with multiple studies on their properties, tolerance, safety and efficacy. However, there are no studies that analyze the effects of consuming these beverages and their interaction with the intestinal microbiota.

Therefore, in addition, it is intended to evaluate the changes in the microbiota, through analysis of stool samples, during the sustained consumption of the beverages under study.

DETAILED DESCRIPTION:
The clinical study has a randomized, double-blind, placebo-controlled design, in which the investigators want to evaluate and compare the effect of hydrating drink A, hydrating drink B, and hydrating drink C (placebo).

Hydration drink A. Water with electrolytes and glucose Hydration drink B. Water with electrolytes and calorie-free sweetener Hydrating drink C. Water with coloring and flavoring. placebo product

625ml containers, administered during sports practice in several intakes according to protocol. Total fluid intake will be 625 ml per training session, 3 times/week over a 4-week period

During the study, each volunteer will make 3 visits: visit 1 (before starting the consumption of the product), visit 2 or 1st control and visit 3 or 2nd control, at the end of the study.

Recruitment or initial interview (Visit 1/Week 0)

In order to recruit volunteers, all interested subjects who meet the criteria below will be informed in detail about the study. Knowing in detail the characteristics of the study and the implications of their participation, the volunteers will be able to sign the informed consent if participants so wish. Before signing, volunteers will have ample time to review and consider the detailed information and ask the researcher questions if participants wish. The volunteer recruitment process will continue until the desired sample size is reached.

Once the informed consent has been signed, a physician trained for the study will carry out the initial interview where it is verified that the subject meets all the inclusion criteria and none of the exclusion criteria, as well as her clinical history.

The investigator will assign the participant the next participant number in the study and, according to a previously prepared randomization list, the treatment that will be received during the study will be assigned.

At this initial visit, a physical examination will be performed that will include weight, height, body mass index (BMI), blood pressure, and heart rate. In addition, the volunteer will take a sample of peripheral blood, urine and feces.

The value of perceived effort will be recorded according to the Borg CR-10 Scale in the last session of high-intensity aerobic exercise performed.

Sufficient treatment will be provided for the entire study and the method of administration will be indicated.

Prior hydration instructions will be indicated (consumption of 500 ml of water during the 2 hours prior to the exercise session) for the control visits in weeks 2 and 4, with the aim that all participants attend in a fit state. optimal hydration.

In this way, clinical baseline values will be obtained to be compared during follow-up visits.

Exercise Session 1 (Visit 2/Week 2) Prior to the start of the session, the investigators will ensure that the volunteer has followed the hydration instructions given at the initial visit.

In this second session, the first control will be carried out, coinciding with 2 weeks from the start of taking the product. In it, the training and hydration protocol will be applied using the different drinks under study and the Borg perceived exertion scale will be passed at the end of the exercise session.

A measurement of body weight will be made before and after the physical exercise session.

Between 30 and 60 minutes after the exercise routine, a peripheral blood sample will be taken. At 90 minutes, a urine sample will be collected. During the time elapsed between the end of the exercise session and the taking of samples, the volunteers will not be able to ingest food or drink. After 90 minutes and all the necessary samples have been taken, the participants will be able to drink and eat on demand.

Exercise session 2. Final Visit (Visit 3/Week 4) The final visit will coincide with the end of the treatment and follow-up period.

The same procedures will be carried out as in visit 2, but in this one, a stool sample will also be collected.

The exercise sessions will be carried out under similar conditions: room, time of practice, temperature and humidity. These sessions will be controlled by the research staff and carried out by staff trained in training.

These will follow the typical structure of high intensity aerobic training sessions, within the different disciplines that follow this methodology in fitness.

In addition to complying with the premises in terms of typology, methodology, structure and general times (established in the training protocol), the control sessions in week 2 and 4 will be exactly the same in relation to the specific design of the exercises and the times .

ELIGIBILITY:
Inclusion Criteria:

* Healthy trained athletes, between 18 and 65 years old, who practice high-intensity aerobic exercise between 3 and 5 times a week
* Signature of the informed consent
* Commitment in terms of compliance with data collection prior to the start of the study, hydration instructions prior to controlled exercise sessions and how to use the product

Exclusion Criteria:

* Chronic disease that, in the opinion of the investigator, contraindicates participation in the study
* Body Mass Index greater than 30
* Acute illness in the last 3 months that has required treatment with steroids
* Medical treatment or nutritional supplement that, in the opinion of the investigator, may interfere with the parameters under study
* Drug use or mild alcoholism (daily consumption >20 g of alcohol in women and > 40 g in men)
* Consumption of antibiotics and/or probiotics in the last 15 days
* Serious allergic diseases
* Inability to communicate with the investigator
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with changes in blood parameters of hydration and recovery: Complete Blood Count | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in complete blood count parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Sodium (mEq/L) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood sodium parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Potassium (mEq/L) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood potassium parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Chlorine (mEq/L) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood chlorine parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Creatine kinase (mg/dL) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood creatine kinase parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Aldolase (U/L) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood aldolase parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Lactate (mg/dL) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood lactate parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Osmolality (mOsm/Kg) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood osmolality parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: AST (U/L) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood AST parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Urea (mg/dL) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood urea parameters at weeks 2 and 4
Number and percentage of participants with changes in blood parameters of hydration and recovery: Creatinine (mg/dL) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session.
  Changes in blood creatinine parameters at weeks 2 and 4

SECONDARY OUTCOMES:
Number and percentage of participants with changes in urinary hydration parameters: Urine osmolality (mOsm/kg) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined 90 minutes after the exercise session.
  Changes in urine osmolality parameters at weeks 2 and 4
Number and percentage of participants with changes in the Borg Scale CR-10 score | At week 0 [T0], the baseline value of the last session of high-intensity aerobic exercise prior to the initial visit will be determined. In week 2 [T1] and 4 [T2] the values will be determined at the end of the exercise session.
  Changes in the Borg Scale of perceived exertion CR-10 score at weeks 2 and 4. Scores on this scale range from 0 to 10 from lowest to highest perceived exertion.
Number and percentage of participants with changes in blood glucose parameters (mg/dL) | At week 0 [T0] the fasting baseline value will be determined. In week 2 [T1] and 4 [T2] the values will be determined between 30 and 60 minutes after the exercise session
  Changes in blood glucose parameters at weeks 2 and 4.
Number and percentage of participants with body mass index changes (BMI) | Baseline fasting weight at week 0 [T0]. Weight before and after exercise sessions at week 2 [T1] and 4 [T2]
  BMI in kg/m^2 changes at weeks 2 and 4. Weight and height will be combined to report BMI in kg/m^2.
Number and percentage of participants with changes in their microbiota composition, alpha diversity and beta diversity, by sequencing the R16s gene of a stool sample | Initial sample collection at week 0 [T0] and final at week 4 [T2]
  Changes in alpha diversity, beta diversity and microbiota composition at week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo MiBioPath. Univesidad Católica San Antonio de Murcia, Guadalupe, Murcia, Spain